CLINICAL TRIAL: NCT07348939
Title: Effect Of Kinesiology Tape On Pain, Posture, Balance And Respiration In Ankylosing Spondylitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Busra Gokgun, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-KAEK-25 2023/03-16
Record Dates: First submitted 2025-12-14; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Ankylosing Spondylitis
Keywords: Ankylosing Spondylitis; Kinesio Taping; Exercise
MeSH Terms: conditions — Spondylitis, Ankylosing; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Patients will be randomly assigned to two groups using a random number table; the first group will receive a home exercise program (ROM, spinal extensor strengthening, posture, balance, and breathing exercises), while the second group will receive both the home exercise program and kinesio taping.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio Tape(Group1) (Experimental): The first group will receive both a home exercise program (ROM, spinal extensor strengthening, posture, balance and breathing exercises) and kinesio taping.
  Interventions: Procedure: Kinesio Taping; Procedure: Exercise
- Exercise(Group 2) (Active Comparator): The second group consists only of a home exercise program (ROM, spinal extensor strengthening, posture, balance and breathing exercises).
  Interventions: Procedure: Exercise

INTERVENTIONS:
Procedure: Kinesio Taping — Kinesiology tapes were applied when the patient was in forward flexion and shoulders were protracted, using functional correction method. Applied without tension at the adhesion point, without any tension in the first 5 from acromioclavicular joint level and then by applying maximum tension and terminating at the lower boundary of costa. Crossing point of the tapes was arranged to be at the lower 1/3 of scapula medial side. Muscle stimulation technique was used to support diaphragm muscle. Origo was xiphoid process, cartilage of 6th costa and lumbar vertebra and insertio was central tendon. Application was made when the patient was standing, with spine at hyperextension, in inspiration and arms in abduction. Tape was applied by following the lower costa curvature from xiphoid process towards lateral. Symmetrically, kinesiology tape was applied dorsally, starting from T12 level and following lower costa curvature.
  Arms: Kinesio Tape(Group1)
Procedure: Exercise — Conventional exercises (Joint ROM, spinal extensor strengthening, posture, balance and respiratory exercises) were explained verbally to both groups and video demonstrations were shown. Patients exercised five days a week for six week, in three sets, consisting of 10 repetitions per day. Exercise practices of the patients were routinely monitored and the patients were encouraged to continue exercise program and phone calls were made to follow-up exercises.

SUMMARY:
This study will investigate the effects of kinesio taping on pain, posture, balance, and respiration in ankylosing spondylitis, and compare its effects with routine home exercises given to this group.

DETAILED DESCRIPTION:
Patients over 18 years of age with a stable course of ankylosing spondylitis will be included in the study. Patients will be randomly divided into two groups using a random number table. The first group will receive a home exercise program (range of motion[ROM], spinal extensor strengthening, posture, balance, and breathing exercises), while the second group will receive both the home exercise program and kinesio taping. Subsequently, comparisons will be made between the groups using visual analog scale (VAS), ROM (cervical and lumbar), Berg Balance Scale, Bath Ankylosing Spondylitis Disease Activity Index (BASDAI), Bath Ankylosing Spondylitis Functional Index (BASFI), Bath AS Metrology Index (BASMI), Modified Schober test, hand-finger-ground distance, chest expansion, and AS(Ankylosing Spondiliytis) quality of life questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age, who had been diagnosed with ankylosing spondylitis

Exclusion Criteria:

Patients with

* active malignancies
* active cellulitis and any infections,
* open wounds
* deep vein thrombosis
* any chronic pulmonary disease,
* fever of unknown origin
* carotid arterial disease,
* vestibular and orthopedic pathologies, affecting balance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-30 (Actual)

PRIMARY OUTCOMES:
VISUAL ANALOG SCALA | From enrollment to the end of treatment at 6 weeks
  This is a scale used to assess pain. It consists of numbered lines on a horizontal line from 0 to 10. The patient marks the line to indicate the intensity of the pain they feel. 0 corresponds to no pain, and 10 corresponds to the most severe pain.
Spinal Pain | From enrollment to the end of treatment at 6 weeks
  The device consists of numbered boxes on a horizontal line from 0 to 10. The patient marks the boxes to indicate the spinal pain they have felt in the last week. 0 corresponds to no pain, and 10 corresponds to the most severe pain.
Nocturnal Spinal Pain | From enrollment to the end of treatment at 6 weeks
  The system consists of numbered boxes on a horizontal line from 0 to 10. The patient marks the boxes to indicate the nocturnal spinal pain they have felt in the past week. 0 corresponds to no pain, and 10 corresponds to the most severe pain.
Fingertips-Floor Distance | From enrollment to the end of treatment at 6 weeks
  The patient is asked to stand upright and touch the tip of their finger to the ground without bending their knees. If there is a limitation, the distance between the fingertip and the ground is measured and recorded. For men, up to 10 cm is considered normal. For women, it is zero.
Modified Schober Test Score | From enrollment to the end of treatment at 6 weeks
  While the patient is standing, a mark is made 10 cm upwards and 5 cm downwards from this prominence. The distance between the two points is 15 cm. The patient performs maximum flexion of their torso. The distance between the two points is measured. 15 cm is subtracted from the measured distance to find the difference. If the difference is less than 5 cm, the test is positive.
BASDAI Score | From enrollment to the end of treatment at 6 weeks
  This is a disease activity-related scale. It consists of 6 questions. Each question has horizontally numbered boxes from 0 to 10, where 0 means none and 10 means very severe. The patient should answer the questions based on their condition over the past week. The questions cover: weakness/fatigue, neck/back/hip pain, joint pain and swelling, touch and pressure sensitivity, and the severity and duration of morning stiffness. The average of the answers to 2 questions related to morning stiffness is added to the sum of the first 4 questions, and then divided by 5 to obtain a combined score.
BASFI Score | From enrollment to the end of treatment at 6 weeks
  The purpose of this scale is to determine and monitor physical functioning in patients with AS. It consists of 10 questions in total: 8 items related to the patients' functional anatomy (bending, reaching, changing position, standing, turning, and climbing stairs) and 2 items assessing the patients' skills related to daily living. The scale is numbered horizontally in rows from 0 to 10, where 0 means easy and 10 means impossible.
BASMI Score | From enrollment to the end of treatment at 6 weeks
  BASMI is a scale used to measure axial skeletal mobility in AS patients and to objectively evaluate clinically significant changes in spinal movement. It was first introduced in 1994 as a 2-point scale. A year later, it was adapted as a 10-point scale, and more recently, its current version as a linear marker has been developed and validated through validation studies.72 It consists of 5 items representing clinical measurements of cervical rotation, tragus-to-wall distance, lumbar flexion (modified Schober), spinal lateral flexion, and maximal intermalleolar distance. Each item is scored between 0 and 10 according to separately defined cut-off values. The ranges are defined as cervical rotation (8.5°-85.0°), tragus-to-wall (10 cm-38 cm), lumbar flexion (7.0 cm-0.7 cm), lumbar lateral flexion (1.2 cm-20 cm), and intermalleolar distance (30 cm-120 cm).
AS Health Assessment Questionnaire | From enrollment to the end of treatment at 6 weeks
  This test is used to assess the physical function of an individual with AS. It consists of 20 questions across 8 categories: dressing, lying down, standing up, eating, walking, hygiene, daily tasks, and grasping. Patients should answer the questions considering their performance over the past week. A scoring system from 0 to 3 is used, with 4 options: 0; easily able, 3; unable to do at all. The total score is divided by the number of questions answered to obtain the final value.
Chest Expanison Diameter | From enrollment to the end of treatment at 6 weeks
  The patient is asked to perform maximal inspiration and expiration. During this time, a measurement is taken and recorded at the 4th intercostal space. The difference between these two results, both in centimeters, is calculated to obtain the desired value.
Respiratory Function Test (RFT) | From enrollment to the end of treatment at 6 weeks
  It is a physiological test that measures airflow as a function of the volume of air taken in and exhaled during respiration and time. Today, it is one of the most basic diagnostic methods frequently used in the diagnosis and monitoring of many lung diseases.
  Dynamic Spirometry It is the first step in respiratory function tests. It is used to evaluate ventilatory capacity. The most important cause of impaired ventilatory capacity is airway obstruction. It is evaluated during forced inspiration and expiration. The measured volume is related to time and expressed with volume-time or flow-volume curves.
  FORCED VITAL CAPACITY (FVC): The volume of air expelled with a forced, rapid, and deep expiration after a deep inspiration.
  Normal: FVC = VC(Vital capacity) Airway obstruction: FVC < VC Normally, 75-80% of the volumes are expelled in the first second. It generally reflects the large airways. It is significantly red
Berg Balance Scale | From enrollment to the end of treatment at 6 weeks
  The Berg Balance Scale is a test used to assess functional balance. It was developed in 1989 by Katherine Berg to evaluate balance functions in the elderly. The scale is useful in predicting the risk and consequences of falls, in evaluating rehabilitation in hospitalized patients, and in assessing the length of hospital stay.
  It consists of 14 items for performance evaluation. Each item is scored between 0 and 4 according to the patient's ability to meet the distance and time requirements of the test. A score of 4 indicates the ability to complete the task without assistance. The highest score is 56. Scores between 0 and 20 indicate impaired balance, 21-40 indicate acceptable balance, and 41-56 indicate good balance.

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Yildirim, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 2 years after the publication of results
Access Criteria: The datasets used and/or analysed during the current study are available from the corresponding author on reasonable request.

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT07348939/Prot_SAP_000.pdf
  • Informed Consent Form (2023-03-24): https://cdn.clinicaltrials.gov/large-docs/39/NCT07348939/ICF_001.pdf